CLINICAL TRIAL: NCT02020369
Title: A Phase III Study on the Safety, Pharmacokinetics and Efficacy of Coagulation Factor VIIa (Recombinant) in Congenital Hemophilia A or B Patients With Inhibitors to Factor VIII or IX
Brief Title: Phase III Study of Coagulation FVIIa (Recombinant) in Congenital Hemophilia A or B Patients With Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: rEVO Biologics (Industry)
Collaborators: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RB-FVIIa-006-13
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Hemophilia A With Inhibitors; Hemophilia B With Inhibitors
MeSH Terms: interventions — Factor VII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FVIIa: 75 µg/kg first, then 225 µg/kg (Experimental): Coagulation Factor VIIa (Recombinant): First Intervention (3 months), Second Intervention (3 months), repeat cycle until study completion.
  Interventions: Biological: Coagulation Factor VIIa (Recombinant)
- FVIIa: 225 µg/kg first, then 75 µg/kg (Experimental): Coagulation Factor VIIa (Recombinant): First Intervention (3 months), Second Intervention (3 months), repeat cycle until study completion.
  Interventions: Biological: Coagulation Factor VIIa (Recombinant)

INTERVENTIONS:
Biological: Coagulation Factor VIIa (Recombinant) — A cross over design to assess the efficacy of 2 separate dose regimens (75µg/kg and 225 µg/kg) of Coagulation Factor VIIa (Recombinant) for the treatment of bleeding episodes in hemophilia A or B patients with inhibitors to Factor VIII/IX

SUMMARY:
The purpose of the study is to assess the safety, efficacy and pharmacokinetics of 2 separate dose regimens (75µg/kg and 225 µg/kg) of Coagulation Factor VIIa (Recombinant) for the treatment of bleeding episodes in hemophilia A or B patients with inhibitors to Factor VIII/IX

DETAILED DESCRIPTION:
This was a global, multicenter, Phase III, prospective, open-label, randomized, crossover study. After obtaining informed consent and performance of screening procedures, patients who met all inclusion and exclusion criteria were randomized to one of two treatment regimens as follows:

* 75 µg/kg treatment regimen
* 225 µg/kg treatment regimen

For each treatment regimen there were two phases:

* Phase A (Initial phase)
* Phase B (Treatment phase)

The assigned treatment regimen was the dose administered in Phase A and was the starting dose in Phase B.

ELIGIBILITY:
Inclusion Criteria:

* be male with a diagnosis of congenital hemophilia A and/or B of any severity
* have one of the following:
* a positive inhibitor test Bethesda Unit (BU) ≥ 5 (as confirmed at screening by the institutional lab), OR
* a BU<5 but expected to have a high anamnestic response to FVIII or FIX, as demonstrated from the subject's medical history, precluding the use of Factor VIII or IX products to treat bleedings, OR
* a BU<5 but expected to be refractory to increased dosing of FVIII or FIX, as demonstrated from the subject's medical history, precluding the use of Factor VIII or IX products to treat bleedings
* be 12 years or older, up to and including 75 years of age (NOTE: different age restrictions may apply per local regulation and/or ethical considerations)
* have at least 3 bleeding episodes of any severity in the past 6 months be capable of understanding and willing to comply with the conditions of the protocol
* have read, understood and provided written informed consent (patient and/or parent(s)/legal guardian(s) if <18 years of age)

Exclusion Criteria:

* have any coagulation disorder other than hemophilia A or B
* be immuno-suppressed (i.e., the patient should not be receiving systemic immunosuppressive medication, cluster of differentiation 4 (CD4) counts at screening should be >200/µl)
* have a known allergy or hypersensitivity to rabbits
* have platelet count <100,000/mL
* have had within one month prior to first administration of the study drug in this study a major surgical procedure (e.g. orthopedic, abdominal)
* have received an investigational drug within 30 days of the first study drug administration, or is expected to receive such drug during participation in this study
* have a clinically relevant hepatic (AST and/or alanine aminotransferase (ALT) >3 times the upper limit of normal) and/or renal impairment (creatinine >2 times the upper limit of normal)
* have a history of arterial and/or venous thromboembolic events (such as myocardial infarction, ischemic strokes, transient ischemic attacks, deep venous thrombosis or pulmonary embolism) within 2 years prior to first dose of study drug, or current New York Heart Association (NYHA) functional classification score of stage II -IV
* have an active malignancy (those with non-melanoma skin cancer are allowed)
* have any life-threatening disease or other disease or condition which, according to the investigator's judgment, could imply a potential hazard to the patient, interfere with the trial participation or trial outcome (e.g., a history of non-responsiveness to bypassing products).

Ages: 12 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Francois Schved, MD, Principal Investigator — Saint Eloi Hospital
Locations (17):
- United States (5):
  - Orthopaedic Hemophilia Treatment Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - University of Colorado Hemophilia and Thrombosis Center, Aurora, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
- Republican Research Center for Radiation Medicine and Human Ecology, Homyel, Belarus
- Specialized Hospital for Active Treatment of Hematological Diseases, Sofia, Bulgaria
- LTD HEMA, Tbilisi, Georgia
- Chaim Sheba Medical Center, Tel-hashomer hospital, Ramat Gan, Israel
- Institute of Hematology and Transfusion Medicine, Warsaw, Poland
- Sandor SRL, Bucharest, Romania
- Russia (3):
  - Kirov Research Institute of Hematology and Blood Transfusion, Kirov
  - Hematology Research Center, Moscow
  - City Outpatient Clinic #37, Saint Petersburg
- Ukraine (2):
  - Kyiv City Clinical Hospital #9, Kyiv
  - Institute of Blood Pathology and Transfusion Medicine of Academy of Medical Sciences of Ukraine, Lviv
- Basingstoke and North Hampshire Hospital, Hemophilia, Hemostasis and Thrombosis Center, Basingstoke, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Young G, Mahlangu J, Boggio LN, Carcao M, Dargaud Y, Escobar M, Giermasz A, Hermans C, Kuriakose P, Miesbach W, Nance D, Rafique A, Sidonio RF Jr, Vilchevska KV, Wang M, Pipe SW. Treatment of severe bleeds with eptacog beta in hemophilia A or B with inhibitors: a post hoc analysis of the PERSEPT 1 and 2 trials. Blood Vessel Thromb Hemost. 2025 Mar 27;2(3):100069. doi: 10.1016/j.bvth.2025.100069. eCollection 2025 Aug. PMID 40765904
- [Derived] Carcao M, Hermans C, Giermasz A, Kessler C, Miesbach W, Quon D, Windyga J, Mahlangu J. Safety and Use of Eptacog Beta 225 microg/kg in Patients With Haemophilia A or B With Inhibitors. Haemophilia. 2025 Sep;31(5):957-965. doi: 10.1111/hae.70083. Epub 2025 Jul 17. PMID 40674256

RESULTS

PARTICIPANT FLOW:
Groups:
- FVIIa: 225 µg/kg First, Then 75 µg/kg: Coagulation Factor VIIa (Recombinant) : First Intervention (3 months), Second Intervention (3 months), repeat sequence for entirety of study.
- FVIIa: 75 µg/kg First, Then 225 µg/kg: Coagulation Factor VIIa (Recombinant): Coagulation Factor VIIa (Recombinant) : First Intervention (3 months), Second Intervention (3 months), repeat sequence for entirety of study.
Period: Overall Study
Arm/Group | FVIIa: 225 µg/kg First, Then 75 µg/kg | FVIIa: 75 µg/kg First, Then 225 µg/kg
Started | 14 | 13
Completed | 11 | 11
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- FVIIa 75 µg/kg First, Then 225 µg/kg; FVIIa 225 µg/kg First, Then 75 µg/kg: Coagulation Factor VIIa (Recombinant): First Intervention (3 months), Second Intervention (3 months), continue cycle until end of study.
- Total: Total of all reporting groups
Arm/Group | FVIIa 75 µg/kg First, Then 225 µg/kg | FVIIa 225 µg/kg First, Then 75 µg/kg | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 3 | 5
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (12.10) | 30.1 (12.98) | 31.0 (12.35)
Sex/Gender, Customized [Number; unit: participants]
  Male (n) | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 12 | 14 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russian Federation | 2 | 3 | 5
  United States | 2 | 2 | 4
  Ukraine | 6 | 6 | 12
  Poland | 1 | 0 | 1
  United Kingdom | 0 | 1 | 1
  Georgia | 1 | 1 | 2
  Bulgaria | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Successfully Treated Mild/Moderate Bleeding Episodes
Description: For the primary efficacy endpoint, successful treatment of a bleeding episode was defined as a combination of the following:
  * "Good" or "Excellent" response noted by the patient
  * Study drug treatment: No further treatment with study drug beyond timepoint for this bleeding episode
  * No other hemostatic treatment needed for this bleeding episode
  * No administration of blood products that would indicate continuation of bleeding beyond timepoint
  * No increase of pain beyond timepoint that could not otherwise be explained
Time Frame: 12 hours after first administration of study drug
Population: Treated Population
Measure: Number (95% Confidence Interval); unit: Proportion of Success of BEs
Units Other Than Participants: Bleeding Episodes (BEs)
Groups:
- FVIIa 75 µg/kg: 75 µg/kg Treatment Regimen at Time of Mild/Moderate Bleeding Episode
- FVIIa 225µg/kg: 225 µg/kg Treatment Regimen at Time of Mild/Moderate Bleeding Episode
Arm/Group | FVIIa 75 µg/kg | FVIIa 225µg/kg
Number analyzed (Participants) | 25 | 25
Number analyzed (Bleeding Episodes (BEs)) | 252 | 213
Proportion of Success of BEs | .849 [.740 to .957] | .932 [.881 to .983]

2. Secondary Outcome: Proportion of Mild/Moderate Bleeding Episodes With Patient (Pt)-Reported "Good" or "Excellent" Responses at 12 Hours
Description: Based on Patient-Reported "Good" or "Excellent" responses as per the below descriptions:
  Good: Symptoms of bleed (e.g., swelling, tenderness, and decreased range of motion in the case of musculoskeletal haemorrhage) had largely been reduced by the treatment, but had not completely disappeared. Symptoms had improved enough to not require more infusions of the study drug.
  Excellent: Full relief of pain and cessation of objective signs of bleed (e.g., swelling, tenderness, and decreased range of motion in the case of musculoskeletal haemorrhage). No additional infusion of study drug was required.
Time Frame: at 12 hours
Population: Treated Population
Measure: Number (95% Confidence Interval); unit: Pt-reported proportion success of BEs
Units Other Than Participants: Bleeding Episodes (BEs)
Groups:
- FVIIa: 75 µg/kg: 75 µg/kg Treatment Regimen at Time of Mild/Moderate Bleeding Episode
- FVIIa: 225 µg/kg: 225 µg/kg Treatment Regimen at Time of Mild/Moderate Bleeding Episode
Arm/Group | FVIIa: 75 µg/kg | FVIIa: 225 µg/kg
Number analyzed (Participants) | 25 | 25
Number analyzed (Bleeding Episodes (BEs)) | 252 | 213
Pt-reported proportion success of BEs | 0.857 [0.750 to 0.964] | 0.937 [0.888 to 0.986]

3. Secondary Outcome: Time to Assessment of a "Good" or "Excellent" Response of Mild/Moderate Bleeding Episodes by the Patient
Description: Categories of Response to Treatment are Described as Follows:
  None: No noticeable effect of the treatment on the bleed or worsening of patient's condition. Continuation of treatment with the study drug was needed.
  Moderate: Some effect of the treatment on the bleed was noticed, e.g., pain decreased or bleeding signs improved, but bleed continued and required continued treatment with the study drug. Good: Symptoms of bleed (e.g., swelling, tenderness, and decreased range of motion in the case of musculoskeletal haemorrhage) had largely been reduced by the treatment, but had not completely disappeared. Symptoms had improved enough to not require more infusions of the study drug.
  Excellent: Full relief of pain and cessation of objective signs of bleed (e.g., swelling, tenderness, and decreased range of motion in the case of musculoskeletal haemorrhage). No additional infusion of study drug was required.
Time Frame: Within 24 hours of Bleeding Episode
Population: Treated Population with non-missing measurements
Measure: Median (95% Confidence Interval); unit: Hours
Units Other Than Participants: Bleeding Episodes with event
Arm/Group | FVIIa: 75 µg/kg | FVIIa: 225 µg/kg
Number analyzed (Participants) | 25 | 25
Number analyzed (Bleeding Episodes with event) | 240 | 208
Hours | 5.98 [5.95 to 6.00] | 3.00 [NA to NA] — The confidence interval (CI) for the median time is a pointwise CI. The median was 3 hours and approximately 30% of bleeding episodes had good/excellent response exactly at 3 hours which made the confidence limits non-calculable.

4. Secondary Outcome: Number of Administrations of Study Drug Per Mild/Moderate Bleeding Episode
Time Frame: Within 24 hours of Bleeding Episode
Population: Treated Population with non-missing measurements
Measure: Mean (Standard Deviation); unit: Number of Administrations of Study Drug
Units Other Than Participants: Bleeding episodes
Groups:
- Factor VIIa: 75 µg/kg: 75 µg/kg Treatment Regimen at Time of Mild/Moderate Bleeding Episode
Arm/Group | Factor VIIa: 75 µg/kg | FVIIa: 225 µg/kg
Number analyzed (Participants) | 25 | 25
Number analyzed (Bleeding episodes) | 252 | 211
Number of Administrations of Study Drug | 2.5 (1.75) | 1.4 (0.96)

5. Secondary Outcome: Total Amount of Study Drug Administered Per Mild/Moderate Bleeding Episode
Time Frame: Through study completion
Population: Treated Population with non-missing measurements
Measure: Mean (Standard Deviation); unit: µg/kg per bleeding episode
Units Other Than Participants: Bleeding Episodes
Arm/Group | FVIIa: 75 µg/kg | FVIIa: 225 µg/kg
Number analyzed (Participants) | 25 | 25
Number analyzed (Bleeding Episodes) | 251 | 211
µg/kg per bleeding episode | 187.868 (131.7982) | 252.963 (78.9732)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected 2 years, 3 months, 2 days
Groups:
- Coagulation Factor VIIa (Recombinant): 75 µg/kg: Coagulation Factor VIIa (Recombinant): 75 µg/kg for 3 months
  Coagulation Factor VIIa (Recombinant): A cross over design to assess the efficacy of 2 separate dose regimens (75µg/kg and 225 µg/kg) of Coagulation Factor VIIa (Recombinant) for the treatment of bleeding episodes in hemophilia A or B patients with inhibitors to Factor VIII/IX
- Coagulation Factor VIIa (Recombinant): 225 µg/kg: Coagulation Factor VIIa (Recombinant) : 225 µg/kg for 3 months
  Coagulation Factor VIIa (Recombinant): A cross over design to assess the efficacy of 2 separate dose regimens (75µg/kg and 225 µg/kg) of Coagulation Factor VIIa (Recombinant) for the treatment of bleeding episodes in hemophilia A or B patients with inhibitors to Factor VIII/IX
Arm/Group | Coagulation Factor VIIa (Recombinant): 75 µg/kg | Coagulation Factor VIIa (Recombinant): 225 µg/kg
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/25
Other Adverse Events (participants affected / at risk) | 3/25 | 3/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coagulation Factor VIIa (Recombinant): 75 µg/kg (N=25) | Coagulation Factor VIIa (Recombinant): 225 µg/kg (N=25)
acute tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
subarachnoid hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coagulation Factor VIIa (Recombinant): 75 µg/kg (N=25) | Coagulation Factor VIIa (Recombinant): 225 µg/kg (N=25)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less